CLINICAL TRIAL: NCT02782507
Title: Cognitive Therapy for Distressing Visual Hallucinations: A Pilot Study
Status: Completed | Type: Observational
Sponsor: Newcastle University (Other)
Collaborators: Northumberland, Tyne and Wear NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: FSF 2010 / 11
Record Dates: First submitted 2013-06-19; First posted 2016-05-25 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Visual Hallucinations; Psychotic Disorders
Keywords: pilot study; CBT trial
MeSH Terms: conditions — Hallucinations; Psychotic Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: CBT for Distressing visual hallucinations — Eight to ten sessions of manualised CBT for distressing visual hallucinations based on existing treatment manuals (ie. Kingdon & Turkington, 2004, Morrison et al., 2005), delivered over 8 to 12 weeks by CBT therapists.
  Subjects will continue to receive treatment as usual throughout the therapy period and will receive appropriate prescription of medication if requested or clinically indicated.
  Other Names: Cognitive Behavioural therapy for visual hallucinations

SUMMARY:
The study is a pilot study of Cognitive therapy for people with psychosis who have distressing visual hallucinations. The aim is to evaluate whether this is an acceptable, feasible and effective treatment. This is a pilot study and there is no randomisation to either CBT or treatment as usual (TAU). If a participant is allocated to the cognitive therapy plus TAU condition then the participant will meet with a therapist on initially a weekly basis and receive up to 8 sessions of CBT over a 2 month period. The participant will also have regular assessments conducted by a researcher who is independent to the treatment group. It is predicted that those people receiving CBT will improve on measures of symptoms, and particularly for measures of visual hallucinations.

DETAILED DESCRIPTION:
Cognitive behavioural therapy (CBT) has been proven to be effective in helping people with distressing psychotic symptoms such as auditory hallucinations or upsetting delusional beliefs. While the majority of hallucinations reported in psychotic disorders are auditory, visual hallucinations (VH) have been reported in 16%-72% of people with psychotic disorders like schizophrenia and schizoaffective disorder. VH appear to be associated with particularly high levels of distress, and impairment. The global severity of illness was significantly higher in people with schizophrenia and VH, as compared to those people without VH. Whilst antipsychotic medication is the first line of treatment for psychotic symptoms like VH, there is evidence that many service users choose to refuse or discontinue their pharmacological treatment. For example, the largest trial to compare atypical antipsychotics found that 74% of patients with a diagnosis of schizophrenia discontinued their medication over 18 months. Hence, there is a need to develop a range of effective treatments. Despite its value in treating auditory hallucinations, at present there is no specific CBT treatment for VH.

We developed a cognitive behavioural model for visual hallucinations. This model has been tested in a recent study of 15 people with psychosis and distressing visual hallucinations which found that it was not the presence of the visual experience per se that led to the distress but the appraisal of it (as being a threat to psychological or physical wellbeing). Such appraisals are targeted in CBT for auditory hallucinations.

The aim of this research is to assess the value of a manualised cognitive behavioural intervention for distressing visual hallucinations by establishing if it reduces distress and disability. The aim is to determine the acceptability of the treatment package, feasibility of recruitment, the ability to deliver the treatment manual as intended, retention in the treatment, a preliminary estimate of effect size and maintenance of any gains at a brief follow up.

ELIGIBILITY:
Inclusion Criteria:

* Meet entry criteria for Early Intervention in Psychosis (EIP) services
* Distressing visual hallucinations
* Age 18-38 years (the usual upper range of the EIP services)

Exclusion Criteria:

* Organic brain disease including dementia, epileptic psychosis, head injury (may be alternative cause of symptoms, or impair cognitive function and ability to do CBT)
* Primary diagnosis of drug or alcohol misuse (as above)
* Impaired intellect severe enough to interfere with ratings (as above)
* In-patient/acute psychiatric care needed at baseline assessment (patients must be well enough to engage in out-patient CBT)
* Previous CBT for psychosis (those previously exposed to the CBT model may be more likely to respond to CBT)

Ages: 18 Years to 38 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: People in Early Intervention in Psychosis services who are reporting distressing visual hallucinations in the past month.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in distress of visual hallucinations as assessed by the Psychotic symptoms rating scale for hallucinations (PSYRATS). | change pre to post intervention which will be on average 3 months
  The PSYRATS measures distress, conviction and preoccupation and impact of life of symptoms such as voices or delusions. It has been adapted to be relevant to visual hallucinations.

SECONDARY OUTCOMES:
Change from baseline on measure of depression (Beck Depression Inventory) | Baseline and at three months
  The BDI is a short, reliable, widely used measure of depression/low mood. It is a self report measure and participants will be asked to complete it before and after the intervention
Change from baseline on measure of symptoms of psychosis as measured by he Schizophrenia Change Scale (SCS). The SCS is a subscale of the Comprehensive Psychopathological Rating Scale (CPRS), (Montgomery, Taylor, & Montgomery, 1978) | baseline and at three months
  The SCS is a short, reliable, widely used measure of symptoms of psychosis. It is a interview based measure and participants will be asked to complete it before and after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Robert Dudley, Ph.D, Principal Investigator — Newcastle University
Locations (1):
- Early Intervention in Psychosis service, Sunderland, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The findings are shared with the individual participants and an anonymised version of the material is to be submitted for publication. The participants have consented to the sharing of anonymised material in this format.